CLINICAL TRIAL: NCT06723249
Title: The Effect of Stingless Bee Honey on BDNF, Oxidative Stress, Depressive Symptoms and Verbal Learning and Memory in Major Depressive Disorders: A Randomized Clinical Trial
Brief Title: Stingless Bee Honey Augmentation in Major Depressive Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Ong Wailoon, Student of Master of science in medical physiology, Hospital Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: USM/JEPeM/KK/24020180; TCTR20240621001 (Registry Identifier: Thai Clinical Trials Registry)
Record Dates: First submitted 2024-12-04; First posted 2024-12-09 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-05

CONDITIONS: Major Depressive Disorder (MDD)
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): The participants under intervention group will receive stingless bee honey. At the same time, they will continue treatment as usual, their pharmacological like antidepressants or psychotherapy
  Interventions: Dietary Supplement: stingless bee honey
- Control group (No Intervention): The participants in the control group will not receive stingless bee honey. They will continue treatment as usual, their pharmacological like antidepressants or psychotherapy

INTERVENTIONS:
Dietary Supplement: stingless bee honey — Participants under intervention group will receive 20g of stingless bee honey in a packet form but participants under control group will not receive any stingless bee honey
  Arms: Intervention group

SUMMARY:
The goal of this clinical trial is to learn if stingless bee honey can be an augmentation supplement in Major Depressive Disorder (MDD) in adults. It will also learn about the adverse effects of the honey. The main questions it aims to answer are:

1. Is there any effect of SBH on depressive symptoms between intervention and control groups in MDD?
2. Are there any effects of SBH on BDNF between intervention and control groups in MDD?
3. Are there any effects of SBH on oxidative stress between intervention and control groups in MDD?
4. Are there any effects of SBH on verbal learning and memory between intervention and control groups in MDD?

There is no placebo.

Participants will:

Take stingless bee honey or nothing every day for 2 months Visit the clinic once every 4 weeks for checkups and tests Report adherence and adverse effects of stingless bee honey on a self-reported online questionnaires

ELIGIBILITY:
Inclusion Criteria:

* Adults with ages 18 to 65
* with Major Depressive Disorder with scores of Beck Depression Inventory Malay version equal or more than 11

Exclusion Criteria:

* Women in pregnancy or breast-feeding.
* Patients who with honey allergy or stingless bee honey allergy.
* Currently taking honey not limited to stingless bee honey or taken honey not limited to stingless bee honey in the past one month.
* comorbidity either with generalized anxiety disorder,
* panic disorder,
* social anxiety disorder,
* bipolar disorder,
* substance-use disorder,
* suicidal ideation or attempt,
* dementia,
* Alzheimer disease,
* diabetic,
* hypertension,
* chronic kidney disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2024-12-15 (Actual); Primary Completion 2025-08-10 (Actual); Study Completion 2025-08-10 (Actual)

PRIMARY OUTCOMES:
Depressive symptoms | Before intervention, at week 4 during the intervention, at week 8 of the intervention
  Depressive symptoms will be assessed using Beck Depression Inventory Malay-version questionnaire, For total score, no depression (1 - 10); mild to moderate (11 -20); moderate to severe (21 - 30); severe (31 - 40); very severe (41 - 63).

SECONDARY OUTCOMES:
Oxidative stress | Before intervention, at week 4 during the intervention, at week 8 of the intervention
  Serum malondialdehyde concentrations in blood will be assessed
Brain derived neurotrophic factors, BDNF | Before intervention, at week 4 during the intervention, at week 8 of the intervention
  Serum BDNF concentrations of blood will be assessed
Verbal learning and memory | Before intervention, at week 4 during the intervention, at week 8 of the intervention
  Verbal learning and memory will be assessed using Malay version of auditory verbal learning test. The highest of total learning (sum of A1-A5 trial) is 75 score which one words = 1 score and the highest for delayed memory (A7 trial) is 15 score
Serum Interleukin-6 | Before intervention, at week 4 during the intervention, at week 8 of the intervention
  Serum IL-6 concentrations of blood will be measured using Elisa kit

CONTACTS AND LOCATIONS:
Overall Officials: Sharifah Zubaidiah, Study Director — Universiti Sains Malaysia; Mohd Zulkifli Mustafa, Study Director — Universiti Sains Malaysia
Locations (1):
- Hospital Universiti Sains Malaysia, Kubang Kerian, Kelantan, Malaysia

IPD SHARING:
Plan to Share IPD: Yes
Raw unprocessed data, without any identifier that could identify patients as individual person such as demographics chacteristics, baseline, week 4 and week 8 primary and secondary outcomes will be shared upon request by others